CLINICAL TRIAL: NCT07010900
Title: Platelet-Rich Plasma Injections From Cord Blood + Penile Traction vs. Penile Traction Alone in Patients With Peyronie's Disease.
Brief Title: Platelet-Rich Plasma Injections From Cord Blood + Penile Traction vs. Penile Traction Alone in Patients With Peyronie's Disease. Open-label, Single-center Randomized Study
Acronym: CB-PRP-TRAC1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB-PRP-TRAC1
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Peyronie Disease; Penile Curvature; PRP Injection; Cord Blood; Randomised Clinical Trial; Penile Injection Therapy
Keywords: penile exteder; peyronie disease; prp; cord blood prp
MeSH Terms: conditions — Penile Induration; Insomnia, Fatal Familial | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penile extender (No Intervention): routine treatment with medical device
- CB-PRP Injection (Experimental): experimental arm
  Interventions: Procedure: Injection

INTERVENTIONS:
Procedure: Injection — patients randomized in intervention group will use also penile extender
  Other Names: CB-PRP
  Arms: CB-PRP Injection

SUMMARY:
The goal of this clinical trial is to learn if Platelet-Rich Plasma Injections from Cord Blood (CB-PRP) is useful in Peyronie disease.

The primary goal is evaluation of patient satisfaction at 1 and 3 months after treatment completion using the PDQ Questionnaire

Secondary Objectives are:

* Measurement of penile curvature measured with a goniometer with spontaneous erection before and after treatment (1 and 3 months)
* Measurement of penile length in stretching before and after treatment (1 and 3 months)
* Evaluation of the improvement in quality of life, through the Short-Form Health Survey 12 (SF-12) health status questionnaire and through the Hospital Anxiety and Depression Scale (HADS)

Participants will be randomized in two groups:

* penile extender alone
* penile extender + CB PRP injection (1 injection every 15 days - 3 in totalinjections)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Peyronie's Disease (IPP) Penile curvature greater than 30 degrees (autophotography in erection with goniometer measurement) Patients candidates for penile traction Age: 18-75 years Good health conditions Preserved erection (IIEF >20) Complete blood count with differential and coagulation within the normal range (platelets between 150,000 and 450,000 μL) HIV, HCV, and HbsAg negative The fertile partner of the patient randomized to the experimental group must use an acceptable highly effective contraceptive method (oral contraceptives, intrauterine device, abstinence, vasectomized partner) for the entire duration of the study Informed consent to the study

Exclusion Criteria:

Coagulopathies, platelet disorders Major active infections Previous penile surgery (excluding circumcision and condyloma removal) Previous infiltrative therapy or penile traction treatment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | From enrollment to the end of follow-up at 6 months
  using PDQ questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chung E, De Young L, Solomon M, Brock GB. Peyronie's disease and mechanotransduction: an in vitro analysis of the cellular changes to Peyronie's disease in a cell-culture strain system. J Sex Med. 2013 May;10(5):1259-67. doi: 10.1111/jsm.12082. Epub 2013 Feb 19. PMID 23421851
- [Result] Almsaoud NA, Safar O, Alshahrani ST, Alwadai R, Alkhaldi SM, Almurayyi M, Alrweili HH, Assiri HM, Al Jubran A, Hakami B, Alzahrani MA. The effect of penile traction device in men with Peyronie's disease on penile curvature, penile length, and erectile dysfunction: a systematic review and meta-analysis. Transl Androl Urol. 2023 Nov 30;12(11):1673-1685. doi: 10.21037/tau-23-310. Epub 2023 Nov 9. PMID 38106680
- [Result] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694
- [Result] Marcovici, I. PRP and Correction of Penile Curvature (Peyronie's Disease). Am J Cosm Surg, 2018. 36: 117.
- [Result] Usta MF, Ipekci T. Penile traction therapy for Peyronie's disease-what's the evidence? Transl Androl Urol. 2016 Jun;5(3):303-9. doi: 10.21037/tau.2016.03.25. PMID 27298777
- [Result] Smith JF, Walsh TJ, Conti SL, Turek P, Lue T. Risk factors for emotional and relationship problems in Peyronie's disease. J Sex Med. 2008 Sep;5(9):2179-84. doi: 10.1111/j.1743-6109.2008.00949.x. Epub 2008 Jul 14. PMID 18638001
- [Result] Gelbard MK, Dorey F, James K. The natural history of Peyronie's disease. J Urol. 1990 Dec;144(6):1376-9. doi: 10.1016/s0022-5347(17)39746-x. PMID 2231932
- [Result] Taylor FL, Levine LA. Peyronie's Disease. Urol Clin North Am. 2007 Nov;34(4):517-34, vi. doi: 10.1016/j.ucl.2007.08.017. PMID 17983892